CLINICAL TRIAL: NCT03865784
Title: Kinesiotape® and Core Exercises in the Improvement of Nonspecific Lumbar Pain, Trunk Flexion, Resistance of the Spinal Erector Musculature and Effort Perception in Federated Boxers
Brief Title: Kinesiotape and Core Exercises in Federated Boxers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Investigación en Hemofilia y Fisioterapia (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: COREKT
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Low Back Pain
Keywords: Boxing; Injuries; Physiotherapy; Kinesiotape; Core; Low back pain
MeSH Terms: conditions — Low Back Pain; Wounds and Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Each session will be held in a group and will last 35 minutes, taking place 2 sessions a week, in a period of 4 weeks. The intervention will be carried out at the end of the training session and after drying the sweat of the area to be treated. After the training, the Core and Kinesiotape exercises with tension and stretching will be performed
  Interventions: Other: Experimental
- Control (Active Comparator): Each session will be held in a group and will last 35 minutes, taking place 2 sessions a week, in a period of 4 weeks. The intervention will be carried out at the end of the training session and after drying the sweat of the area to be treated. After the training, the Core and Kinesiotape exercises technique will be performed without tension or stretching
  Interventions: Other: Control

INTERVENTIONS:
Other: Experimental — The intervention through Core exercises will consist in the application of a protocol of four Core stabilization exercises. This protocol will consist of the following exercises: abdominal plate, bilateral plate, hunting dog and gluteal bridge. The intervention by Kinesiotape will be performed with the subject in a sitting position with both arms relaxed throughout the body, while the physiotherapist will place the bases of the strips without tension, on the sacroiliac joint. Once this is done, proceed to ask the subject to lean forward applying the rest of the strip, except the distal edge, with a tension of between 15 and 25%, finally requesting the subject to rejoin straining the distal base without tension, on the twelfth dorsal spinous process.
  Arms: Experimental
Other: Control — The intervention through Core exercises will consist in the application of a protocol of four Core stabilization exercises. The objective of the application of the technique based on this type of exercise is to improve muscle strength, endurance and neuromuscular control. This protocol will consist of the following exercises: abdominal plate, bilateral plate, hunting dog and gluteal bridge. The intervention by Kinesiotape will be performed with the subject in a sitting position with both arms relaxed throughout the body, while the physiotherapist will place the bases of the strips without tension, on the sacroiliac joint. Once this is done the tape will be placed without tension and sn movement of the subject.
  Arms: Control

SUMMARY:
Introduction. Nonspecific lumbar pain is a very common cause of sports decline in boxers, possibly due to the repetitive movements of flexion and rotation in their sport, so the investigators believe it is interesting to seek an intervention that helps these athletes to reduce their incidence.

Aim. To improve non-specific low back pain, range of motion of trunk flexion; the muscular resistance of the spinal erectors and the subjective perception of the effort in federated boxers older than 18 years.

Study design. Randomized, multicentric and double-blind clinical trial with follow-up period.

Methods. 60 federated boxers of legal age will be recruited, who will be randomly assigned to the study groups: experimental (Core and Kinesiotape® exercises) and control (Core exercises and Kinesiotape® tubes without tension). The intervention will last 4 weeks, with 2 weekly sessions, lasting 35 minutes. Three evaluations will be carried out (pre-treatment, post-treatment and follow-up) for the dependent variables. The analysis of normality will be carried out with the Kolmogorov Smirnov test and in case of homogeneity of the sample, with the t-student test of related samples and the ANOVA of repeated means, the difference between the evaluations and the intra e effect will be calculated. intersubject, respectively.

Expected results. It is expected to observe the effectiveness of the Core and Kinesiotape® exercises in the perception of nonspecific lumbar pain, the range of movement of trunk flexion and lumbar resistance, and the perception of effort.

ELIGIBILITY:
Inclusion Criteria:

* Federated boxers
* Over 18 years
* Male
* With non-specific back pain that does not incapacitate them for the realization of their sport or work activity.

Exclusion Criteria:

* Federated boxers with lumbar injury with medical diagnosis
* Who are or have been treated by pharmacological or physiotherapy in the last 6 months
* Presenting allergies or alterations of the skin
* Not sign the informed consent document.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-04-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline pain perception after treatment and at month: VAS | Screening visit, within the first seven days after treatment and after one month follow-up visit
  Pain perception measurement will be measured with the visual analogue scale, which is represented by a line from 0 mm to 100 mm indicating at the ends the states of 'no pain '(0) and' as much pain as it can bear' (10) . The EVA scale is measured as the distance between the line of 'no pain 'and that marked by the subject. A change greater than 13 mm between the two would be considered clinically relevant

SECONDARY OUTCOMES:
Change from baseline pain perception at the pressure after treatment and at month: pressure algometer | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The perception of pain at the pressure will be calculated with a pressure algometer (model Baselin de Quirumed), whose assessment varies from 0 to 10 kg. It consists of a rubber block of 1 cm2, performing the evaluation by applying pressure in the paravertebral area to the height of the 3rd and 4th lumbar spinous processes, with the subject in the prone position. The unit of measure is kg. the subject indicating the perception of pain by means of an acoustic signal (for example: "stop"). The greater the units of measurement (kg), the better the perception of the subject's pain.
Change from baseline perception of effort after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  To measure the perception of effort, the Borg scale will be used. This measuring instrument is designed to linearly describe exercise intensity and heart rate. In the simplest version of this scale, the numbers from 0 to 10 are used. The number 0 indicates a non-existent perception of the effort, and the number 10 implies an extremely strong perception of the intensity of the effort.
Change from baseline trunk flexion after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The trunk flexion will be evaluated by applying the Schober test. A mark will be made at the lumbosacral junction, and two other marks on the skin (one at 10 cm above the lumbosacral junction and another at 5 cm below). The subjects should flex their trunk to the maximum without flexing the knees and at the same time measure the distance between the upper and lower marks. The unit of measurement of this test is in centimeters, where a higher score indicates a greater range of trunk movement in flexion.
Change from baseline trunk flexion after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The trunk flexion will be evaluated the finger-ground test. The subject will stand in an anthropometric box, and perform a trunk flexion with the extended legs stretching both arms towards the ground and facing the palms towards their legs. The subjects must maintain that position for two seconds until the measurement is taken. The unit of measurement of this test is in centimeters, where a higher score indicates a greater range of trunk movement in flexion.
Change from baseline resistance of the lumbar extensor musculature after treatment and at month | Screening visit, within the first seven days after treatment and after one month follow-up visit
  The resistance of the lumbar extensor musculature will be evaluated through the Biering Sorensen test. This test consists of placing the subject in a prone position with the lower limbs fixed to the stretcher and the upper part of the body extended from the hip to the head, towards the outside of the stretcher. You will be asked to hold the horizontal position with your arms crossed over your chest as long as possible. This test has by unit of measurement the time (in seconds), where at higher valuation, greater resistance of the extensor musculature.

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Comunity of Madrid, Spain